CLINICAL TRIAL: NCT03814733
Title: A Phase 1, Randomized, Double-blind, Double-dummy, Placebo-controlled, 5-period, Crossover Study Assessing the Effects of Rapastinel Compared to Alprazolam, Ketamine, and Placebo on Simulated Driving Performance in Normal Healthy Participants
Brief Title: Assessment of Effect of Rapastinel on Driving Performance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: RAP-PK-18
Record Dates: First submitted 2018-11-15; First posted 2019-01-24 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Driving Performance
MeSH Terms: interventions — GLYX-13 peptide; Alprazolam; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Rapastinel High Dose (Experimental): Participants will be administered single IV doses of rapastinel, ketamine, rapastinel matched placebo, and ketamine matched placebo, and single oral doses of alprazolam and alprazolam matched placebo in a randomized crossover manner.
  Interventions: Drug: Rapastinel
- Rapastinel Low Dose (Experimental): Participants will be administered single IV doses of rapastinel, ketamine, rapastinel matched placebo, and ketamine matched placebo, and single oral doses of alprazolam and alprazolam matched placebo in a randomized crossover manner.
  Interventions: Drug: Rapastinel
- Alprazolam (Active Comparator): Participants will be administered single IV doses of rapastinel, ketamine, rapastinel matched placebo, and ketamine matched placebo, and single oral doses of alprazolam and alprazolam matched placebo in a randomized crossover manner.
  Interventions: Drug: Alprazolam
- Ketamine (Active Comparator): Participants will be administered single IV doses of rapastinel, ketamine, rapastinel matched placebo, and ketamine matched placebo, and single oral doses of alprazolam and alprazolam matched placebo in a randomized crossover manner.
  Interventions: Drug: Ketamine
- Placebo for Rapastinel (Placebo Comparator): Participants will be administered single IV doses of rapastinel, ketamine, rapastinel matched placebo, and ketamine matched placebo, and single oral doses of alprazolam and alprazolam matched placebo in a randomized crossover manner.
  Interventions: Drug: Rapastinel Matched Placebo
- Placebo for Alprazolam (Placebo Comparator): Participants will be administered single IV doses of rapastinel, ketamine, rapastinel matched placebo, and ketamine matched placebo, and single oral doses of alprazolam and alprazolam matched placebo in a randomized crossover manner.
  Interventions: Drug: Alprazolam Matched Placebo
- Placebo for Ketamine (Placebo Comparator): Participants will be administered single IV doses of rapastinel, ketamine, rapastinel matched placebo, and ketamine matched placebo, and single oral doses of alprazolam and alprazolam matched placebo in a randomized crossover manner.
  Interventions: Drug: Ketamine Matched Placebo

INTERVENTIONS:
Drug: Rapastinel — Participants will be administered single IV doses of rapastinel, ketamine, rapastinel matched placebo, and ketamine matched placebo, and single oral doses of alprazolam and alprazolam matched placebo in a randomized crossover manner.
  Arms: Rapastinel High Dose; Rapastinel Low Dose
Drug: Alprazolam — Participants will be administered single IV doses of rapastinel, ketamine, rapastinel matched placebo, and ketamine matched placebo, and single oral doses of alprazolam and alprazolam matched placebo in a randomized crossover manner.
  Arms: Alprazolam
Drug: Ketamine — Participants will be administered single IV doses of rapastinel, ketamine, rapastinel matched placebo, and ketamine matched placebo, and single oral doses of alprazolam and alprazolam matched placebo in a randomized crossover manner.
  Arms: Ketamine
Drug: Rapastinel Matched Placebo — Participants will be administered single IV doses of rapastinel, ketamine, rapastinel matched placebo, and ketamine matched placebo, and single oral doses of alprazolam and alprazolam matched placebo in a randomized crossover manner.
  Arms: Placebo for Rapastinel
Drug: Alprazolam Matched Placebo — Participants will be administered single IV doses of rapastinel, ketamine, rapastinel matched placebo, and ketamine matched placebo, and single oral doses of alprazolam and alprazolam matched placebo in a randomized crossover manner.
  Arms: Placebo for Alprazolam
Drug: Ketamine Matched Placebo — Participants will be administered single IV doses of rapastinel, ketamine, rapastinel matched placebo, and ketamine matched placebo, and single oral doses of alprazolam and alprazolam matched placebo in a randomized crossover manner.
  Arms: Placebo for Ketamine

SUMMARY:
Based on the pharmacological class of rapastinel, this study will be conducted to evaluate the participant's driving performance after single IV doses of rapastinel as compared with single oral doses of alprazolam, a benzodiazepine that demonstrates driving impairment, and placebo in healthy participants.

ELIGIBILITY:
Inclusion Criteria

* Participant possesses a valid driver's license and is an active driver. Drives a minimum of 5,000 miles (about 8,000 km) per year for the previous 3 years.
* Participant has a regular sleep pattern, is not engaged in shift-work, and in general, has at least 7 hours of sleep each night (bedtime occurs between 21:00 and 24:00 hours).

Exclusion Criteria

* A history within 2 years of, or current intervention for, a sleeping disorder (including excessive snoring, obstructive sleep apnea) or a chronic painful condition that interferes with the participant's sleep.
* A history of difficulty in falling asleep or staying asleep in the previous 3 months that is considered clinically significant by the investigator.
* Participant has traveled across 1 or more time zones (transmeridian travel) in the 14 days before study intervention or is expected to travel across 1 or more time zones during the study.
* Expected to work on a rotating shift during their participation in the study.
* Participant works a night shift.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Simulated driving performance as measured by SDLP using the CRCDS-MiniSim for rapastinel compared with placebo and positive control (alprazolam) | Day 1 of each intervention

SECONDARY OUTCOMES:
simulated driving performance as measured by SDLP using the CRCDS-MiniSim for rapastinel compared with a clinical comparator (ketamine) | Day 1 of each intervention
Karolinska Sleepiness Scale (KSS) | Day 1 of each intervention
  The KSS is a participant self-reported measure of situational sleepiness and provides an assessment of alertness/sleepiness. The KSS is a 9-point categorical scale, where 1 = "extremely alert" and 9 = "extremely sleepy-fighting sleep".
Self-perceived safety to drive ("Right now do you feel safe to drive?) | Day 1 of each intervention
Visual Analog Scale to assess participant's motivation and self-appraisal of their driving performance | Day 1 of each intervention
CogScreen SDC Test | Day 1 of each intervention
Proportion of abnormal lane exceedance events | Day 1 of each intervention
Average Speed (mph) | Day 1 of each intervention
Total collisions | Day 1 of each intervention
Number of exceeded cornering speed threshold events | Day 1 of each intervention
Divided attention: average number of correct responses | Day 1 of each intervention
  Participants are asked to answer periodic questions during the driving simulation.
Divided attention: average number of errors | Day 1 of each intervention
  Participants are asked to answer periodic questions during the driving simulation.
Divided attention: average reaction time | Day 1 of each intervention
Rapastinel blood plasma concentration | Day 1 of each intervention
Adverse Events | Up to 66 days
Proportion of abnormal electrocardiograms | Up to 66 days
Columbia-Suicide Severity Rating Scale | Up to 66 days
  The C-SSRS is a clinician-ratedinstrument that reports theseverity of both suicidal ideation and behavior. Suicidal ideation is classified on a 5-item scale: 1 (least severe) to 5 (most severe).

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Fang Su, Study Director — Allergan
Locations (2):
- Collaborative Neuroscience Network, San Clemente, California, United States
- Algorithme Pharma, Aurora, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Su S, Kay G, Hochadel T, Rojo J, Christopher Stein J, Boinpally R, Periclou A. A randomized, multicenter trial assessing the effects of rapastinel compared to ketamine, alprazolam, and placebo on simulated driving performance. Clin Transl Sci. 2022 Jan;15(1):255-266. doi: 10.1111/cts.13145. Epub 2021 Nov 7. PMID 34423904